CLINICAL TRIAL: NCT05321160
Title: Comparison of Esketamine Versus Sevoflurane Add to Dexmedetomidine-based Sedation for Minor Ophthalmology Procedure in Children: A Randomized Controlled Trial.
Brief Title: Comparison of the Sedation Effect of Esketamine and Sevoflurane for Pediatric Ophthalmological Procedure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EA and esketamine
Record Dates: First submitted 2022-03-25; First posted 2022-04-11 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Adverse Event
Keywords: adverse event; sevoflurane; esketamine
MeSH Terms: interventions — Esketamine; Ketamine; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group E (Experimental): 1ug· kg-1 dexmedetomidine and 0.01mg·kg-1 atropine was administered intravenously. 0.25mg·kg-1 esketamine was administered by vein in one minute, and 0.25mg·kg-1 esketamine was given at the beginning of the surgery.
  Interventions: Drug: Esketamine
- Group S (Active Comparator): 1ug· kg-1 dexmedetomidine and 0.01mg·kg-1 atropine was administered intravenously. 4% sevoflurane(FIO2=100%, 3L·min-1) was used to induce anesthesia by mask inhalation and 2-4 % sevoflurane (adjusted according to the depth of the anaesthesia,FIO2=100%, 2L·min-1) was maintained.
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Esketamine — 0.25 mg/kg esketamine for induction and 0.25 mg/kg esketamine at the beginning of surgery
  Other Names: s(+)ketamine
  Arms: Group E
Drug: Sevoflurane — 4% sevoflurane for induction and 2-4% sevoflurane for maintain
  Other Names: Sevoflurane Inhalation Solution
  Arms: Group S

SUMMARY:
Emergence agitation is the most common reason for post-anesthesia care unit delay. Sevoflurane is used frequently inhalational anaesthetic agent to provide pediatric anaesthesia because of the nonirritant nature. It has been successfully used for keeping spontaneous breathing without tracheal intubation. However, sevoflurane may cause emergence agitation as the incidence varied from 10%-80%. Although there are many sedative agents to reduce its incidence, such as propofol, midazolam, a2 adrenergic receptor agonists and ketamine, the efficacy remains limited.

Ketamine, a neuroleptic anesthetic agent, contains two optical isomers, s(+)-ketamine (esketamine) and R(-)-ketamine. Esketamine is a right-handed split of ketamine, which has enhanced analgesic potency and lower incidence of psychotropic side effects compared to ketamine. It stimulate breathing due to N-Methyl-D-Aspartate receptor blockade, and could even effectively countered remifentanil-induced respiratory depression. The investigators compared the effectiveness of esketamine and sevoflurane in reducing the incidence of emergence agitation after painless ophthalmological procedure in pediatric patients.

DETAILED DESCRIPTION:
Ophthalmological procedure such as suture remove, intraocular pressure (IOP) measurement, slit-lamp and fundoscopy are most frequently performed in operation with minor surgical stimulus, and the the duration of surgery is very short. Several anesthestic agents are available,but it is hard to balance short effect and fast rotation in post-anesthesia care unit. Emergence agitation is the most common reason for post-anesthesia care unit delay. Sevoflurane is used frequently inhalational anaesthetic agent to provide pediatric anaesthesia because of the nonirritant nature. It has been successfully used for keeping spontaneous breathing without tracheal intubation. However, sevoflurane may cause emergence agitation as the incidence varied from 10%-80%. Although there are many sedative agents to reduce its incidence, such as propofol, midazolam, a2 adrenergic receptor agonists and ketamine, the efficacy remains limited.

Ketamine, a neuroleptic anesthetic agent, contains two optical isomers, s(+)-ketamine (esketamine) and R(-)-ketamine. Esketamine is a right-handed split of ketamine, which has enhanced analgesic potency and lower incidence of psychotropic side effects compared to ketamine. It stimulate breathing due to N-Methyl-D-Aspartate receptor blockade, and could even effectively countered remifentanil-induced respiratory depression. Additionally, several studies have reported ketamine could reduced agitation, but there is no study about esketamine on emergence agitation. The investigators compared the effectiveness of esketamine and sevoflurane in reducing the incidence of emergence agitation after painless ophthalmological procedure in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists physical status 1-2
* required to remove the stitches by microscope after corneal surgeries

Exclusion Criteria:

* psychiatric disorders
* cardiovascular disorders
* glaucoma
* contraindications to nasal intubation

Ages: 3 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 116 (Actual)
Dates: Start 2022-03-28 (Actual); Primary Completion 2023-05-14 (Actual); Study Completion 2023-05-17 (Actual)

PRIMARY OUTCOMES:
the incidence of respiratory depression | duration from the time patient received induction to the time of leaving to the ward, average 1 hour
  respiratory rate <12 times per min or weak chest undulation
the incidence of desaturation | duration from the time patient received induction to the time of leaving to the ward, average 1 hour
  the incidence of oxygen saturation below 95% caused by anesthetic agent.
the incidence of hypotension | duration from the time patient received induction to the end of the anesthesia, average 15 minutes.
  the incidence of systolic blood pressure< 30% of basal systolic blood pressure and lasted >5 minutes.
the incidence of hypertension | duration from the time patient received induction to the end of the anesthesia, average 15 minutes.
  the incidence of systolic blood pressure > 30% of basal systolic blood pressure
the incidence of tachycardia | duration from the time patient received induction to the end of the anesthesia, average 15 minutes.
  the incidence of heart rate increase over 30% of pre-induction and>120 beats per minute.
the incidence of bradycardia | duration from the time patient received induction to the end of the anesthesia, average 15 minutes.
  the incidence of heart rate less than 60 beats per minute
the incidence of emergence agitation | duration from the time patients arrived the post-anesthesia care unit to the time of leaving to the ward, average 20 minutes
  the incidence of emergence agitation

SECONDARY OUTCOMES:
length of stay in the post-anesthesia care unit | duration from the time patients arrived the post-anesthesia care unit to the time of leaving to the ward, average 20 minutes
  the time of patients staying in post-anesthesia care unit
CPS score | scores at the time point of 1 minutes after extubation
  The Cole 5-point scale CPS) score included five behaviors: 1=sleeping; 1=awake,calm;3=irritable, crying;4=inconsolable crying; 5=severe restlessness, disorientation.
intraocular pressure | the time after intubation and topical anesthesia within 1 minute
  intraocular pressure after induction
diastolic pressure | 1minutes before induction; 1minutes before intubation; 1minutes after intubation; 3 minutes after intubation
  diastolic pressure
systolic pressure | 1minutes before induction; 1minutes before intubation; 1minutes after intubation; 3 minutes after intubation
  systolic pressure
heart rate | 1minutes before induction; 1minutes before intubation;1minutes after intubation,3 minutes after intubation
  heart rate
extubation time | duration from the time that patients arrived in post-anesthesia care unit to the time of extubation, average 10 minutes
  extubation time

CONTACTS AND LOCATIONS:
Overall Officials: Fang Tan, Principal Investigator — Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University
Locations (1):
- Anesthesiology Department of Affiliated Eye and ENT Hospital, Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Liao R, Li JY, Liu GY. Comparison of sevoflurane volatile induction/maintenance anaesthesia and propofol-remifentanil total intravenous anaesthesia for rigid bronchoscopy under spontaneous breathing for tracheal/bronchial foreign body removal in children. Eur J Anaesthesiol. 2010 Nov;27(11):930-4. doi: 10.1097/EJA.0b013e32833d69ad. PMID 20683333
- [Background] Cravero J, Surgenor S, Whalen K. Emergence agitation in paediatric patients after sevoflurane anaesthesia and no surgery: a comparison with halothane. Paediatr Anaesth. 2000;10(4):419-24. doi: 10.1046/j.1460-9592.2000.00560.x. PMID 10886700
- [Background] Welborn LG, Hannallah RS, Norden JM, Ruttimann UE, Callan CM. Comparison of emergence and recovery characteristics of sevoflurane, desflurane, and halothane in pediatric ambulatory patients. Anesth Analg. 1996 Nov;83(5):917-20. doi: 10.1097/00000539-199611000-00005. PMID 8895263
- [Background] White PF, Schuttler J, Shafer A, Stanski DR, Horai Y, Trevor AJ. Comparative pharmacology of the ketamine isomers. Studies in volunteers. Br J Anaesth. 1985 Feb;57(2):197-203. doi: 10.1093/bja/57.2.197. PMID 3970799
- [Background] Patrizi A, Picard N, Simon AJ, Gunner G, Centofante E, Andrews NA, Fagiolini M. Chronic Administration of the N-Methyl-D-Aspartate Receptor Antagonist Ketamine Improves Rett Syndrome Phenotype. Biol Psychiatry. 2016 May 1;79(9):755-764. doi: 10.1016/j.biopsych.2015.08.018. Epub 2015 Aug 24. PMID 26410354
- [Background] Eich C, Verhagen-Henning S, Roessler M, Cremer F, Cremer S, Strack M, Russo SG. Low-dose S-ketamine added to propofol anesthesia for magnetic resonance imaging in children is safe and ensures faster recovery--a prospective evaluation. Paediatr Anaesth. 2011 Feb;21(2):176-8. doi: 10.1111/j.1460-9592.2010.03489.x. No abstract available. PMID 21210891